CLINICAL TRIAL: NCT02982382
Title: Neurophysiological and Functional Effects of Manipulative Therapy and Pain Education in Individuals With Chronic Nonspecific Low Back Pain
Brief Title: Effects of Manipulative Therapy and Pain Education in Individuals With CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Catarina Federal University (Other)
Responsible Party: Principal Investigator, Clecio Vier, Principal Investigator, Santa Catarina Federal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cvier; U1111-1190-4899 (Other: World Health Organization - WHO)
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Musculoskeletal Manipulations; Neurophysiology; Education
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Manipulation, Spinal; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Manipulative Treatment (Experimental): Subjects will receive Manipulative Therapy
  Interventions: Other: Manipulative Therapy; Other: Pain Education
- Pain Education (Sham Comparator): Subjects will receive Pain Education and manual contact over lumbar region
  Interventions: Other: Pain Education; Other: Sham

INTERVENTIONS:
Other: Manipulative Therapy — Subjects will receive techniques of High Velocity and Low Amplitude (HVLA) or grade V manipulation to the lumbar region (lumbar roll), and pain education based on the biopsychosocial approach.
  Other Names: Manual Therapy; Grade V Manipulation; Spinal Manipulation
  Arms: Manipulative Treatment
Other: Pain Education — Individuals will receive pain education based in a biopsychosocial approach
  Other Names: Neuroscience Pain Education
Other: Sham — The individuals will receive a simulation of spinal manipulation (sham) involving manual contact over lumbar region totaling 5 minutes.
  Arms: Pain Education

SUMMARY:
The burden of low back pain more than doubled in the last 20 years, probably caused by biopsychosocial factors. Some noninvasive treatments have been applied in individuals with chronic nonspecific low back pain as spinal manipulation and pain education. However, it is not already clear the neurophysiological effects of these treatments.The purpose of this research is to verify the effects of the technique of spinal manipulation and pain education in individuals with chronic low back pain

DETAILED DESCRIPTION:
The outcomes will be subjective pain (measured by Numeric Pain Rating Scale), pressure pain threshold (measured by Algometer), disability (measured by Roland-Morris Disability Questionnaire), fear and avoidance beliefs (measured by Fear Avoidance Beliefs Questionnaire), risk of poor prognosis (measured by STarT Back Screening Tool), quality of life (measured by Short Form-12v2) and blood biomarkers (measured by ELISA). The data will be collected by a blinded assessor.

Individuals eligibility is going to be assessed by blinded assessor to determine if they are or not eligible for this research. Then, they will be informed about the objectives of this study and asked to sign the consent form. Afterward, the sociodemographic data will be recorded. The data related to the research outcomes will be collected by the blinded assessor at baseline assessment, after six weeks and three months.

Random Allocation Before the treatment begins, one of the researchers not involved in the recruiting and assessment will allocate the individuals in one of the groups. Block randomization will be used; it is going to generate by randomization.com, this site will create a list with the randomization sequence, which will be only seen by the physical therapists that will treat the individuals.

Statistical Methods

Sample size calculation The sample size calculation was calculated with the A-priori test with the following specifications: Statistical test ANCOVA, the effect size of 0.25, the statistical power of 80%, and an alpha level of 5%. As a result, the study requires a sample size of 64 per group or 128 individuals in total.

Analysis of effects of treatment Our research will use the intention-to-treat principles. The descriptive data and the scores of RMDQ, SBST, FABQ, SF-12v2 and NPRS as well as the pressure pain threshold means and the values of inflammatory biomarkers, before and after interventions, will be tabbed on Microsoft Excel 2010. To see the effect of treatment is going to be used statistical based on intention-to-treat principles, statistical analyses will be used to analyses data of individuals socio-demographics and clinics characteristics, and they will be presented by mean and standard deviation. To compare the groups, Shapiro-Wilk test will be applied to test the normality distribution of data, depending on this distribution will be used ANOVA one-way for parametric data or Kruskal-Wallis test for non-parametric data. To compare groups on the pre-intervention period another ANOVA-one way or another Kruskal-Wallis will be applied.

Covariance analysis (ANCOVA) will be conducted to assess the effect of treatment on the following outcomes: Scores obtained on RMDQ, FABQ, SF-12v2, SBST and NPRS, pressure pain threshold and the blood biomarkers concentrations, utilizing the post-treatment means as dependent variables, the pre-treatment means as co-variables and the group as fixed factor.

To the relationships among the variables must be applied the Pearson correlation coefficient to parametric data and Spearman correlation coefficient to nonparametric data. To classify the relationships will be used the Munro's classification, where values between 0.26 and 0.49 will be low, values between 0.50 and 0.69 will be moderate, between 0.70 and 0.89 will be high values, and between 0.90 and 1.0 will be considered very high. For all of these analyses will be used the Statistical Package for the Social Sciences (IBM SPSS version 20.0, IBM Corp, Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* Chronic episodes of nonspecific LBP for at least six months
* Pain on movement for at least one direction (flexion, extension, side bending or rotation of the trunk)
* At least score 3 in NPRS.

Exclusion Criteria:

* 1) Previous history of lumbar myelopathy, rheumatic disease, tumors, peripheral or central neurological disorders
* 2) Historical of trauma, fracture or surgery in lumbar region;
* 3) Nerve root compression signs: important muscle weakness affecting lower limb, decrease or abolish of patellar and calcaneus reflex and decrease of dermatomes sensibility of lower limbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks after randomization
  Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Pain Intensity | Baseline, 6 weeks and 3 months
  Numeric Pain Rating Scale (NPRS)
Disabilty | baseline, 6 weeks and 3 months
  Rolland Morris Disability Questionnaire (RMDQ)
Pressure Pain Threshold | Baseline, 6 weeks and 3 months
  The pressure pain threshold will be assessed by algometer. It will be realized three times in each point (Five centimeters of the right and left side of the spinal process of L1, L3 and L5, and on the muscle belly of tibialis anterior).
Fear and Beliefs about pain | Baseline, 6 weeks and 3 months
  Fear Avoidance Belief Questionnaire (FABQ)
Risk of poor prognosis | Baseline, 6 weeks and 3 months
  STarT Back Screening Tool (SBST)
Quality of Life | Baseline, 6 weeks and 3 months
  Short-Form Health Survey 12 version 2 (SF-12v2)
Serum Level of Cytokines | Baseline, 6 weeks
  Enzyme Linked Immunosorbent Assay (ELISA) to TNF-α, IL-1β, IL-4, IL-6, IL-8, IL-12, IL-10, IL-15, MIP-4, CCL18, MCP-3 / CCL7, MCP-2 / CCL8, IGP - 10 / CXCL10, Stromal Lymphopoietin Receptor (TSLR), Interferon Gamma and CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Clécio Vier, PhD Student, Principal Investigator — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Florianópolis, Santa Catarina, Brazil